CLINICAL TRIAL: NCT03745157
Title: A Prospective Non-interventional Study Investigating the Treatment Effect of Switching From Insulin Glargine to Ryzodeg® (Insulin Degludec/Insulin Aspart) in a Real World Adult Population With Type 2 Diabetes in Japan
Brief Title: RESILIENT: A Research Study, Looking at How Ryzodeg® Works in People With Type 2 Diabetes in Local Clinical Practice in Japan
Acronym: RESILIENT
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN5401-4441; U1111-1208-5143 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-11-14; First posted 2018-11-19 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Type 2 Diabetes requiring insulin therapy: Patients with type 2 diabetes requiring insulin therapy in Japanese routine clinical practice previously treated with insulin glargine (IGlar)
  Interventions: Drug: Insulin Degludec/Insulin Aspart

INTERVENTIONS:
Drug: Insulin Degludec/Insulin Aspart — Patients will be treated with commercially available Insulin Degludec/Insulin Aspart (Ryzodeg®) in a pre-filled pen injector (FlexTouch®) according to routine clinical practice at the discretion of the treating physician in accordance with the Ryzodeg® label in Japan

SUMMARY:
The purpose of the study is to collect information on how Ryzodeg® works in real world participants. Participants will get Ryzodeg® as prescribed to them by the study doctor. The study will last for about 6 to 8 months. The participants will be asked questions about their health and their diabetes treatment as part of their normal study doctor's appointment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures related to recording of data according to the protocol
* The decision to initiate treatment with commercially available insulin Ryzodeg® has been made by the patient/legally acceptable representative and the treating physician before and independently from the decision to include the patient in this study
* Male or female, age more than or equal to 20 years (the legal age of adulthood) at the time of signing informed consent
* Diagnosed with type 2 diabetes (T2D) for at least 26 weeks prior to signing informed consent
* Available and documented glycosylated haemoglobin (HbA1c) value less than or equal to 12 weeks prior to initiation of Ryzodeg® treatment
* For at least 26 weeks prior to initiation of Ryzodeg® treatment, one of the following must apply: A) Treated with insulin glargine (IGlar) (any formulation, including biosimilar IGlar). B) Treated with IGlar (any formulation, including biosimilar IGlar) and IGlar U300 for at least 12 weeks prior to initiation of Ryzodeg®

Exclusion Criteria:

* Previous participation in this study. Participation is defined as signed informed consent.
* Pregnancy
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Hypersensitivity to Ryzodeg® or to any of the excipients
* Previously treated with Ryzodeg®

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes requiring insulin therapy
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
Change in local laboratory measured glycosylated haemoglobin (HbA1c) | From baseline (up to 12 weeks prior to treatment initiation (week 0)) to end of study visit or at discontunuation (-2 to +8 weeks at 26 weeks)
  Measured in %point

SECONDARY OUTCOMES:
Change in total insulin dose | From baseline (the most recent dose prior to treatment initiation (week 0)) to end of study visit or at discontinuation (-2 to +8 weeks at 26 weeks)
  Measured in units/day
Change in basal insulin dose | From baseline (the most recent dose prior to treatment initiation (week 0)) to end of study visit or at discontinuation (-2 to +8 weeks at 26 weeks)
  Measured in units/day
Change in prandial insulin dose | From baseline (the most recent dose prior to treatment initiation (week 0)) to end of study visit or at discontinuation (-2 to +8 weeks at 26 weeks)
  Measured in units/day
Change in local laboratory measured fasting plasma glucose (FPG) | From baseline (up to 12 weeks prior to treatment initiation (week 0)) to end of study (-2 to +8 weeks at 26 weeks)
  Measured in mg/dL
The incidence of patient recollection of non-severe hypoglycaemic episodes | Pre- and post initiation of treatment with Ryzodeg®. Episodes occurring within 4 weeks prior to initiation of treatment with Ryzodeg® and within 4 weeks prior to end of study visit or at discontinuation (-2 to +8 weeks at 26 weeks)
  Measured in episodes/person-year
The incidence of patient recollection of nocturnal non-severe hypoglycaemic episodes | Pre- and post initiation of treatment with Ryzodeg®. Episodes occurring within 4 weeks prior to initiation of treatment with Ryzodeg® and within 4 weeks prior to end of study visit or at discontinuation (-2 to +8 weeks at 26 weeks)
  Measured in episodes/person-year
The incidence of patient recollection of overall severe hypoglycaemic episodes | Pre- and post initiation of treatment with Ryzodeg®. Episodes occurring within 26 weeks prior to initiation of treatment with Ryzodeg® and within 26 weeks prior to end of study visit or at discontinuation (-2 to +8 weeks at 26 weeks)
  Measured in episodes/person-year
The incidence of patient recollection of nocturnal severe hypoglycaemic episodes | Pre- and post initiation of treatment with Ryzodeg®. Episodes occurring within 26 weeks prior to initiation of treatment with Ryzodeg® and within 26 weeks prior to end of study visit or at discontinuation (-2 to +8 weeks at 26 weeks)
  Measured in episodes/person-year
Change in selected patient reported outcomes: Diabetes Therapy Related Quality of Life (DTR-QoL) | From baseline to end of study visit or at discontinuation (-2 to +8 weeks at 26 weeks). Baseline defined as visit 1 (week 0)
  Score (on a scale from 0-100, where 100 is the highest health related quality of life (HRQoL))

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (26):
- Japan (26):
  - Novo Nordisk Investigational Site, Arakawa-ku, Tokyo
  - Novo Nordisk Investigational Site, Chuo-ku, Tokyo
  - Novo Nordisk Investigational Site, Fukuoka-shi, Fukuoka
  - Novo Nordisk Investigational Site, Fukushima
  - Novo Nordisk Investigational Site, Higashiosaka-shi, Osaka
  - Novo Nordisk Investigational Site, Hokkaido
  - Novo Nordisk Investigational Site, Hosu-gun, Ishikawa
  - Novo Nordisk Investigational Site, Kanagawa
  - Novo Nordisk Investigational Site, Kawagoe-shi, Saitama
  - Novo Nordisk Investigational Site, Kawaguchi-shi, Saitama
  - Novo Nordisk Investigational Site, Kisarazu-shi, Chiba
  - Novo Nordisk Investigational Site, Kita-ku, Tokyo
  - Novo Nordisk Investigational Site, Nagano
  - Novo Nordisk Investigational Site, Saitama-shi, Saitama
  - Novo Nordisk Investigational Site, Sapporo-shi, Hokkaido
  - Novo Nordisk Investigational Site, Sendai-shi, Miyagi
  - Novo Nordisk Investigational Site, Shimotsuga-gun, Tochigi
  - Novo Nordisk Investigational Site, Shimotsuke-shi, Tochigi
  - Novo Nordisk Investigational Site, Shinjuku-ku, Tokyo
  - Novo Nordisk Investigational Site, Shizuoka-city, Shizuoka
  - Novo Nordisk Investigational Site, Shizuoka-shi, Shizuoka
  - Novo Nordisk Investigational Site, Tochigi
  - Novo Nordisk Investigational Site, Tokyo
  - Novo Nordisk Investigational Site, Tsuchiura-shi,Ibaraki
  - Novo Nordisk Investigational Site, Yaizu-shi, Shizuoka
  - Novo Nordisk Investigational Site, Yokohama-shi, Kanagawa

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Shigiyama F, Liu L, Nordahl H, Suzuki R, Yamamoto Y, Hirose T. A Real-World, Prospective, Non-interventional Study of Adults with T2D Switching to IDegAsp from Glargine U100 or U300 in Japan. Diabetes Ther. 2021 Sep;12(9):2405-2421. doi: 10.1007/s13300-021-01117-8. Epub 2021 Jul 25. PMID 34304385